CLINICAL TRIAL: NCT07223320
Title: Feasibility and Preliminary Effectiveness of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) + Functional Strength Training (FST) in Children With Spinal Muscular Atrophy (SMA): a Pilot Study
Brief Title: HABIT-ILE + FST in Children With SMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-429
Record Dates: First submitted 2025-09-25; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: SMA - Spinal Muscular Atrophy
Keywords: HABIT-ILE; Functional strength training; Pediatric; Rehabilitation; Motor control; Intensive
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined HABIT-ILE + FST (Experimental): Participants receive a combined intervention consisting of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) and Functional Strength Training (FST). Both components are delivered as an integrated, intensive motor learning-based program aimed at improving upper and lower limb function in children with SMA .Subject will participate in a HABIT-ILE + FST camp format for 6 hours/day, one day/week for 15 weeks.
  Interventions: Other: Combined Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) + functional strength training (FST)

INTERVENTIONS:
Other: Combined Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) + functional strength training (FST) — Goal-directed, task-specific training for both the upper and lower extremity, and postural control with targeted strengthening exercises to enhance motor control and facilitate the achievement of functional goals

SUMMARY:
This single-arm pilot study will assess the feasibility and preliminary effectiveness of an intensive motor skill intervention (HABIT-ILE) combined with functional strength training (FST) in children with SMA who are receiving disease-modifying therapies. Participants will attend one 6-hour HABIT-ILE + FST session each weekend (Saturday or Sunday) for 15 weeks, for a total of 90 hours of training. Feasibility will be evaluated through questionnaires, and effectiveness through standardized motor function assessments.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a severe neuromuscular disorder marked by the progressive degeneration of alpha motor neurons in the spinal cord and brainstem, resulting in proximal muscle atrophy and weakness. Based on age of onset and the motor function achieved, children were historically categorized into functional groups. However, recent advances leading to the development of disease-modifying therapies (DMTs) have transformed the management of SMA. Outcomes are now primarily determined by the timing of DMT initiation, with early treatment-ideally before symptom onset-showing significant efficacy in improving motor function and survival. Despite these therapeutic breakthroughs, rehabilitation remains a cornerstone of care for children with SMA. Current clinical guidelines emphasize physical activity, muscle strengthening, and stretching. However, few controlled studies have rigorously evaluated these interventions, and even fewer have examined their combined effects with DMTs. This gap underscores the need for innovative, evidence-based rehabilitation strategies that can complement pharmacological treatments and further promote functional outcomes. Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) is an intervention that integrates bimanual coordination with postural control and gross motor training. Grounded in motor skill learning principles, HABIT-ILE delivers high-intensity, structured practice of progressively increased motor difficulty tasks and functional activities, emphasizing voluntary active movement. The approach has demonstrated efficacy in children aged 6 months to 18 years with cerebral palsy (CP), a non-progressive neurodevelopmental disorder caused by early brain injury. Although SMA and CP differ in pathophysiology, both conditions involve motor impairments that may respond to intensive, task-specific motor training. In individuals with SMA, central neuroplastic mechanisms may help compensate for peripheral motor deficits, while targeted motor training could optimize recruitment and efficiency of residual motor units in the muscle. Strength training, in particular, has demonstrated beneficial effects in individuals with SMA, suggesting that emphasizing skill training requiring increasing endurance and progressively increasing the weights of objects participants handled, may be especially advantageous. In this context, augmenting HABIT-ILE with a functional strength training (FST) component tailored to individual goals may further enhance motor outcomes in this population. The aim of this pilot proposal is to evaluate the feasibility and preliminary efficacy of HABIT-ILE + FST in children with SMA receiving DMTs. Children with SMA will attend one 6-hour HABIT-ILE + FST session each weekend (either Saturday or Sunday) for 15 weeks, adding up to a total of 90 hours. It is hypothesized that this intervention will be well tolerated by children, enhance the acquisition of new motor skills, and foster greater functional independence in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SMA
* Able to participate in all pre and post intervention assessments
* Able to understand and speak English
* Able to understand directions (no significant cognitive delay or serious behavioral issues that would limit participation)
* Receiving a stable dose of disease-modifying therapies for at least 6 months prior to enrollment.

Exclusion Criteria:

* Orthopedic surgery within the last year (confound)
* Initiation of any new pharmaceutical treatment during the study period
* Participation in a clinical trial of an investigational therapy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility questionnaire | Immediately after the intervention
  Feasibility questionnaire completed by both the child and their parents to assess the acceptability of the intervention (including child satisfaction and physical comfort, and parent feedback), as well as its demand and practicality.

SECONDARY OUTCOMES:
Hammersmith Functional Motor Scale -Expanded (HFMSE) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Gross motor function measure; range: 0 to 66; higher scores indicate better motor function
Revised Upper Limb Module (RULM) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Upper limb function measure; range: 0 to 37; higher scores indicate better uper limb function
Endurance Shuttle box and blocks test (ESBBT) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Dexterity and upper extremity endurance/fatigability; range: O to 20 minutes (time to limitation); higher times correspond to better endurance
6-Minute Walk Test (6MWT) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Walking endurance measure; range: 0 meters to the maximim distance the participant can walk in 6 minutes; higher distances reflect better ambulatory function and endurance.
10 Meter Walking Test (10MWT) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Assesses gait speed by recording the time required to walk 10 meters, which is then expressed in meters per second. Scores range from 0 m/s (unable to walk) up to approximately 2 m/s in healthy individuals. Higher walking speed reflects better ambulatory function.
Timed Up and Go (TUG) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Functional mobility and dynamic balance measure. The TUG measures the time required to rise from a chair, walk 3 meters, turn around, return, and sit down. The outcome is expressed in seconds, with lower times reflecting better functional mobility and balance
30-Second Sit-to-Stand Test (30STS) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Lower limb strength and endurance measure; range: 0 (unable to stand) to higher values reflecting better lower limb strength and endurance
Trunk Control Measurement Scale (TCMS) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Static and dynamic trunk control measure; range: 0 to 58 points; higher scores indicating better trunk control
Spinal Muscular Atrophy EFFORT (SMA EFFORT) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Questionnaire of perceived physical fatigability (ages 12 years and older); different subscales; higher scores indicating greater perceived fatigue
Canadian Occupational Performance Measure (COPM) | 4 assessments: Baseline 1, baseline 2 (1 week), post intervention (16 weeks), 3 months follow-up
  Interview of occupational performance and satisfaction; range: 1 to 10 for each item, with higher scores indicating better performance or greater satisfaction.
Daily activity logs | Every day during the intervention (assessed up to 15 weeks)
  Implementation feasibility measure

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cerebral Palsy Research, Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mercuri E, Finkel RS, Muntoni F, Wirth B, Montes J, Main M, Mazzone ES, Vitale M, Snyder B, Quijano-Roy S, Bertini E, Davis RH, Meyer OH, Simonds AK, Schroth MK, Graham RJ, Kirschner J, Iannaccone ST, Crawford TO, Woods S, Qian Y, Sejersen T; SMA Care Group. Diagnosis and management of spinal muscular atrophy: Part 1: Recommendations for diagnosis, rehabilitation, orthopedic and nutritional care. Neuromuscul Disord. 2018 Feb;28(2):103-115. doi: 10.1016/j.nmd.2017.11.005. Epub 2017 Nov 23. PMID 29290580
- [Background] Bleyenheuft Y, Gordon AM. Hand-arm bimanual intensive therapy including lower extremities (HABIT-ILE) for children with cerebral palsy. Phys Occup Ther Pediatr. 2014 Nov;34(4):390-403. doi: 10.3109/01942638.2014.932884. Epub 2014 Oct 1. PMID 25271469
- [Background] Bleyenheuft Y, Ebner-Karestinos D, Surana B, Paradis J, Sidiropoulos A, Renders A, Friel KM, Brandao M, Rameckers E, Gordon AM. Intensive upper- and lower-extremity training for children with bilateral cerebral palsy: a quasi-randomized trial. Dev Med Child Neurol. 2017 Jun;59(6):625-633. doi: 10.1111/dmcn.13379. Epub 2017 Jan 30. PMID 28133725